CLINICAL TRIAL: NCT00308126
Title: Phase IV, Open-Label, Randomized, Albumin-Controlled, Parallel Group, Multicenter Study to Evaluate the Effect of Medium Molecule HES (130/0.4) in Complications for Patients After Abdominal Surgery
Brief Title: Study to Evaluate the Effect of Hydroxyethyl Starch (HES) in Complications of Patients After Abdominal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fresenius Kabi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BFP501
Record Dates: First submitted 2006-03-28; First posted 2006-03-29 (Estimated); Last update posted 2007-12-11 (Estimated); Status verified 2006-03

CONDITIONS: Postoperative Complications
Keywords: Abdominal operation
MeSH Terms: conditions — Postoperative Complications | interventions — Hydroxyethyl Starch Derivatives; HES 130-0.4

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Hydroxyethyl Starch 130/0.4 (Voluven)

SUMMARY:
Purpose: To compare the incidence of post-surgery complications and evaluate relevant parameters within 28 days after an operation in HES (130/0.4) and albumin treated groups

Study Design: Open-label, active controlled, parallel group, randomized, multi-center study. Per protocol, 624 patients required in 6 study centers.

Hypothesis: No difference in rate of postoperative (post-op) complications between HES and albumin groups

DETAILED DESCRIPTION:
Since the application of surgical operations, postoperative complications have been the area surgeons explored the most. Though surgical technological advances make it possible for most patients to recover from an operation, the prevention and management of the postoperative complications are still important for surgeons.

Traditionally, the level of albumin is an important marker for the prognosis of the patient. When the level of albumin is below 35 g/L, the mortality rate and other complications will increase significantly, so albumin has become the widely used colloid liquid in fluid therapy for postoperative patients. Actually, the body cannot utilize exogenous albumin and it takes 6-7 days for the body to synthesize new albumin. There is dispute concerning whether albumin should be used in postoperative treatments for severely ill patients. The well-known SAFE study found there was no difference in the efficacy between albumin and crystalloids for severe patients in the 28-day observation time. A meta analysis of 24 studies involving 1419 patients came to the conclusion that administration of albumin could increase the mortality rate in patients. The high price of albumin is another target for extensive criticism.

On the other hand, maintaining colloid osmotic pressure at a certain level in the circulatory system is essential for postoperative patients to stabilize hemodynamics, reduce tissue edema, improve recovery, so it is beneficial for patients to replace albumin with Voluven (130/0.4). Voluven (130/0.4) is a medium-molecular-weight hydroxyethyl starch produced by Fresenius Kabi Pharmaceutical Co. Ltd, and is widely used clinically in volume replacement therapy. Its efficacy and safety are proved by its clinical practices, however, its effect in patients with postoperative complications is not clear. The study will compare the effect of Voluven (130/0.4) and albumin on the occurrence of postoperative complications in patients with an abdominal operation to provide guidance on selection of safe and economic volume replacement therapy for postoperative patients.

STUDY OBJECTIVES

To compare the effect of Voluven (130/0.4) to that of albumin for occurrence of postoperative complications in patients with abdominal surgery from the day of the operation to 28th day after the operation.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 75, male or female
* After abdominal operation of medium scale or above (including but not limited to: gastric cancer eradication, rectal cancer eradication, hepatic lobectomy, corpus and cauda pancreatectomy)
* Hemoglobin (Hb) no less than 70g/L; serum albumin no less than 30 g/L before operation
* Blood loss during operation no more than 2000 ml

Exclusion Criteria:

* Known to be allergic to HES or albumin
* Urine output less than 500 ml/24 hours
* Intra-cranial hemorrhage
* Liver transplantation
* Use colloid other than study drugs
* Lung edema
* Pregnant, lactating female
* Participate in other clinical study within 30 days
* Poor compliance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 624
Dates: Start 2005-06; Study Completion 2006-09

PRIMARY OUTCOMES:
Occurrence of any postoperative complication stipulated in protocol within 28 days after abdominal operation

SECONDARY OUTCOMES:
28th day after abdominal operation

CONTACTS AND LOCATIONS:
Overall Officials: Yupei Zhao, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College (PUMC) Hospital, Beijing, China